CLINICAL TRIAL: NCT00708487
Title: A Controlled Randomized Trial Evaluating the Effect of Lowered Incubator Oxygen Tension on Live Births in a Predominantly Blastocyst Transfer Program
Brief Title: Live Births With Low Oxygen Blastocyst Culture
Acronym: Oxygen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Health Resources (Other)
Responsible Party: Marius Meintjes, Presbyterian Hospital of Dallas
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PresbyterianHDallasARTSO2
Record Dates: First submitted 2008-06-29; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Infertility; Pregnancy Rate, Live Birth; In Vitro Fertilization
Keywords: in vitro fertilization; oxygen concentration; blastocyst; live birth; embryo
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 5% oxygen embryo culture condition
  Interventions: Other: Embryo incubator oxygen concentration
- 2 (Active Comparator): 21% oxygen embryo culture condition
  Interventions: Other: Embryo incubator oxygen concentration

INTERVENTIONS:
Other: Embryo incubator oxygen concentration — Two concentrations of oxygen are currently used to culture the embryos of infertile patients in commercial human IVF programs - 21% and 5%.

SUMMARY:
The potentially damaging effect of free O2 radicals to cultured embryos may be reduced by adding scavengers to the culture media or by reducing the incubator O2 levels. However, lowering the O2 in the culture environment can be expensive, troublesome and may not be justifiable. The objective of this study is to evaluate the effect of lowered incubator O2 tension on live birth rates in a predominately day-5 embryo transfer program. The hypothesis of this study is that a lowered (more physiological)oxygen concentration in embryo culture incubators will increase live birth rates for in vitro fertilization patients. 230 first-cycle women undergoing routine IVF or ICSI with ejaculated sperm will be randomized in a prospective clinical trial and stratified for patient age and physician. Embryos of patients will be randomly assigned for culture in either a 21% O2 (atmospheric) or 5% O2 (reduced) environment. Clinical endpoints monitored will be rates of implantation, clinical pregnancy, live birth and blastocyst cryopreservation.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to determine if a more physiological oxygen concentration (5%) will improve clinical outcomes when compared with the industry standard of 21%.

Background: For embryos to grow in the incubator, atmospheric gas concentrations should be as close to possible to those seen in the oviduct or uterus. Currently, atmospheric (non-physiological, 21%) oxygen concentrations are used in the incubators to culture the embryos of infertility patients of the Presbyterian ARTS laboratories. Literature suggest that culturing animal embryos in a reduced oxygen environment will significantly improve embryo quality and clinical outcomes. Both 5% and atmospheric oxygen concentrations are routinely used for embryo culture in the human IVF laboratories, however, very few commercial human IVF facilities invest in oxygen control as it is more expensive to maintain and labor intensive to implement. The goal is to use lower oxygen concentrations in the future if clinical improvement justifies the expense and increased labor associated with low oxygen culture.

Project Summary: Study design: The study will be conducted in a prospective, randomized way. Two treatment groups are considered: 1) existing atmospheric oxygen concentration in embryo incubators 2) lower 5% oxygen concentration in embryo culture incubators. To allow for the well-documented decline in pregnancy rates with increased age, patients will be stratified within 4 age groups and 3 physicians within each treatment. The age groups are: donor eggs; <35 years; 35 to 37 years; and 38 to 40 years as determined on the day of egg retrieval.

Endpoints Measured: The endpoints measured will be embryo cryopreservation-biochemical pregnancy-, clinical pregnancy-, ongoing pregnancy-, live birth- and embryo implantation rates.

Number of Patients in the Study: To detect a difference of 10% in pregnancy rates, 150 patients should be included in each treatment group. With the current patient volume, it should take less than one year to complete the study. Differences in implantation rates may be detected earlier (more embryos transferred than patients enrolled). Should significance differences in pregnancy rates become evident before the full number of patients is enrolled, the study may be terminated.

Study Location: The study will be conducted at the ARTS facility of Presbyterian Hospital of Plano.

Criteria for Inclusion of Subjects: All patients undergoing a first IVF cycle or any donor oocyte cycle is eligible to participate in this laboratory comparison. The eggs may be fertilized with conventional IVF methodology or by using intracytoplasmic sperm injection (ICSI). When performing ICSI, ejaculated sperm must be used. Patients using their own eggs must be 40 years of age or younger on the day of egg retrieval. The Presbyterian Hospital ARTS Program performed ~900 egg retrievals in 2000. Of these, ~500 would have met the inclusion criteria of this study.

Criteria for Exclusion of Subjects: To reduce the tremendous patient variability seen in the infertile patient population, only first cycle patients 40 years of age or younger on the day of egg retrieval should participate.

Sources of Research Material: Patients will be enrolled in this study from the regular patient pool presented to the Presbyterian ARTS Program for treatment of infertility. Data will not be collected specifically for research purposes. Data to be used are collected on all ARTS patients, regardless of participation in the study.

Recruitment of Subjects: Subjects for this study will be recruited from the regular patient pool presented to the ARTS Program for the treatment of infertility. Patients that will meet the inclusion criteria of this study can be identified prospectively. Information about the study will be included in the routine, biweekly, group laboratory and nursing orientation sessions.

Potential Risks: Patients consenting to the comparison will allow their embryos to be cultured in either the standard atmospheric oxygen concentration or in a reduced, more physiological oxygen concentration. Atmospheric (21%) oxygen concentrations is the current standard in this program. Both methods are considered industry standard. To our best knowledge and as reported in animal literature, low oxygen culture should do better rather than worse under the conditions proposed for this study. No other culture conditions or culture media compositions/ingredients that will be applied during this comparison is experimental. However, when atmospheric oxygen concentrations and lowered (5%) oxygen concentrations are compared in a controlled, randomized way as suggested in this comparison, the ARTS Program can not guarantee that the pregnancy outcome will be equivalent for both treatment groups. Therefore, by being randomized, a patient may be included in a group with a lower success rate.

Special Precautions: If it should become clear early in the study that either one of the treatments are superior to the other, the study will be discontinued and the best conditions implemented for future patients.

ELIGIBILITY:
Inclusion Criteria:

* First IVF cycle or donor oocyte cycle
* IVF or ICSI
* Ejaculated sperm only for ICSI
* <41 years of age

Exclusion Criteria:

* One or more failed IVF cycles

  * 40 years of age
* Using testicular or epididymal sperm for fertilization

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 1999-08; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Live birth | 9 months

SECONDARY OUTCOMES:
Implantation rate | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marius Meintjes, PhD, Principal Investigator — Texas Health Resources
Locations (1):
- Presbyterian Hospital of Palno, Plano, Texas, United States

REFERENCES:
- [Derived] Meintjes M, Chantilis SJ, Douglas JD, Rodriguez AJ, Guerami AR, Bookout DM, Barnett BD, Madden JD. A controlled randomized trial evaluating the effect of lowered incubator oxygen tension on live births in a predominantly blastocyst transfer program. Hum Reprod. 2009 Feb;24(2):300-7. doi: 10.1093/humrep/den368. Epub 2008 Oct 16. PMID 18927130